CLINICAL TRIAL: NCT07330609
Title: Clinical, Radiographic, and Digital Evaluation of the Effects of Autogenous Grafts Harvested From Different Palatal Sites and Applied During Second-stage Implant Surgery on the Peri-implant Mucosa
Brief Title: Clinical, Radiographic, and Digital Evaluation of the Effects of Autogenous Grafts on Peri-implant Mucosa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ezgi Gürbüz, Associate Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSBU001
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Peri-implant Health; Free Gingival Graft; Peri-implant Mucositis

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial with parallel groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronal palatal tissue (Experimental): Participants in this group will receive grafts including marginal and interdental palatal gingiva.
  Interventions: Procedure: Coronal palatal tissue
- Apical palatal tissue (Active Comparator): Participants in this group will receive grafts harvested from approximately 1.5 mm apical to the palatal gingival margin.
  Interventions: Procedure: Apical palatal tissue

INTERVENTIONS:
Procedure: Coronal palatal tissue — This group will receive palatal grafts including marginal and interdental gingiva. This coronal palatal tissue will be applied to the peri-implant tissue at the second-stage implant surgery.
  Arms: Coronal palatal tissue
Procedure: Apical palatal tissue — This group will receive palatal grafts harvested from approximately 1.5 mm apical to the gingival margin. This graft will be applied to the peri-implant tissue at the second-stage implant surgery.
  Arms: Apical palatal tissue

SUMMARY:
This study aims to evaluate the effects of autogenous grafts harvested from different palatal regions on the peri-implant mucosa when applied during second-stage dental implant surgery.

Clinical, radiographic, and digital assessment methods will be used to investigate the early effects of these grafts on peri-implant mucosal width and thickness. In addition, peri-implant tissue health and patient-reported outcomes will be evaluated to compare the effectiveness of the grafting techniques in peri-implant soft tissue management.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Systemically healthy patients
* Presence of premolar or molar tooth loss in the mandible
* Adequate mesiodistal and interocclusal space for implant and restoration placement
* At least four months elapsed since tooth extraction
* Alveolar bone width of at least 6 mm and sufficient alveolar bone height to allow implant placement without compromising anatomical structures
* Full-mouth plaque and bleeding scores less than 20%
* Presence of opposing teeth in occlusion
* Keratinized mucosa width in the relevant region less than 2 mm
* Keratinized mucosa thickness in the relevant region of 2 mm or less
* Presence of a healthy second premolar in the maxilla
* Provision of written informed consent and permission for the use of data for research purposes

Exclusion Criteria:

* Poor oral hygiene
* Uncontrolled periodontal disease
* Pregnancy or lactation at any stage of the study
* Uncontrolled diabetes mellitus
* Immunocompromised patients
* Previous radiotherapy to the head and neck region
* Diseases or medications affecting bone metabolism
* Antibiotic use within the three months prior to the procedure
* Smoking more than 10 cigarettes per day
* Pre- or simultaneous bone augmentation prior to implant placement
* Lack of primary stability at the time of implant placement

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-08-02 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Peri-implant Mucosal Thickness | Pre-operative and post-operative (before implant placement, 3rd month (second-stage implant surgery), 6th month after implant placement, and 12th month after prosthetic loading)
  The primary outcome is the change in peri-implant mucosal thickness measured at four time points using clinical and digital methods.

SECONDARY OUTCOMES:
Keratinized Mucosa Width | Pre-operative and post-operative (before implant placement, 3rd month (second-stage implant surgery), 6th month after implant placement, and 12th month after prosthetic loading)
  Keratinized tissue width will be measured from the mid-buccal aspect of the edentulous area.
Vestibular Depth | Pre-operative and post-operative (before implant placement, 3rd month (second-stage implant surgery), 6th month after implant placement, and 12th month after prosthetic loading)
  Vestibular depth is defined as the vertical distance between the midcrestal area and the point of greatest concavity of the mucosal fold.
Modified Plaque Index | Postoperative 6th month after implant placement and 12th month after prosthetic loading
  Modified plaque index will be measured at six points around each implant by an index with a minimum value of 0 and a maximum of 3.
Modified Bleeding Index | Postoperative 6th month after implant placement and 12th month after prosthetic loading
  Modified bleeding index will be measured at six points around each implant by an index with a minimum value of 0 and a maximum of 3.
Peri- implant Probing Depth | Postoperative 6th month after implant placement and 12th month after prosthetic loading
  Peri-implant probing depth will be measured at six points around each implant.
Mucosal Recession | 12th month after prosthetic loading
  Mucosal recession will be measured as the distance between the implant abutment interface and the mucosal margin.
Marginal Bone Level | Pre-operative and post-operative (before implant placement, 3rd month (second-stage implant surgery), 6th month after implant placement, and 12th month after prosthetic loading)
  Marginal bone level will be measured on periapical radiographs taken by the parallel technique.
Pink Esthetic Score (PES) | Postoperative 3rd month (second-stage implant surgery) and 12th month after prosthetic loading
  Peri-implant soft tissue esthetics will be evaluated using the Pink Esthetic Score with a minimum value of 0 and a maximum of 14.
Postoperative Pain Assessment | Postoperative 14 days (daily after graft application)
  Postoperative pain as patient-reported outcome will be recorded using a visual analog scale (VAS; 0-100).
Analgesic Consumption | Postoperative 14.days (after graft application)
  The amount of analgesic medication used (mg) will be recorded.
Patient Satisfaction | Postoperative 14.days (after graft application)
  Patient satisfaction with the surgical procedure will be assessed using a three-point Likert scale (0 = no, 1 = maybe, 2 = yes).
Patient-Perceived Esthetic Outcome | 12th month after prosthetic loading
  Patient perception of peri-implant soft tissue esthetics will be evaluated using a visual analog scale (VAS; 0-100).
Oral Health-Related Quality of Life | Postoperative 3rd month (second-stage implant surgery) and 12th month after prosthetic loading
  Oral health-related quality of life will be assessed using the Oral Health Impact Profile (OHIP-14) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zigdon H, Machtei EE. The dimensions of keratinized mucosa around implants affect clinical and immunological parameters. Clin Oral Implants Res. 2008 Apr;19(4):387-92. doi: 10.1111/j.1600-0501.2007.01492.x. Epub 2008 Feb 11. PMID 18266873
- [Background] Bassetti RG, Stahli A, Bassetti MA, Sculean A. Soft tissue augmentation procedures at second-stage surgery: a systematic review. Clin Oral Investig. 2016 Sep;20(7):1369-87. doi: 10.1007/s00784-016-1815-2. Epub 2016 Apr 4. PMID 27041111